CLINICAL TRIAL: NCT00171795
Title: Efficacy and Safety of Rivastigmine in Patients With Traumatic Brain Injury and Cognitive Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CENA713BDE01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury,; cognitive impairment,; rivastigmine
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
This study is designed to investigate the efficacy and safety of rivastigmine compared with placebo in patients with traumatic brain injury and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury confirmed by available brain imaging (CT or MRI) and be at least 52 weeks post injury
* Neuropsychologic disturbances indicated by: impaired memory (reduction of below 1 standard deviation (SD) of the mean on the California Verbal Learning Test (CVLT) and impaired executive function (reduction of below 1 standard deviation (SD) of the mean on the Verbal Memory Learning Test (VLMT) and Tower of London Test (ToL) and impaired attention (reduction of below 1 standard deviation (SD) of the mean on the Test Battery for Attentional Performance (TAP)
* Be required to have had sufficient education to read, write, and effectively communicate
* Be cooperative, able to ingest oral medication, and able to complete all aspects of the study and capable of doing so, either alone or with the aid of a responsible caregiver according to the investigator's judgement

Exclusion Criteria:

* A current diagnosis of cerebrovascular disease, any primary neurodegenerative disorder, or any other causes of neuropsychologic disturbances
* A current diagnosis of active, uncontrolled seizure disorder or major depression, or any other diagnosis that may interfere with the patient's response to study medication
* An advanced, severe or unstable disease of any type that may interfere with efficacy evaluations
* Female patients with child-bearing potential who are breast-feeding, pregnant or not practicing non-hormonal contraception

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-11; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
20 week's treatment with rivastigmine on selective attention compared with placebo in patients with TBI and cognitive impairment

SECONDARY OUTCOMES:
Safety of rivastigmine
Change from baseline to week 20 in cognitive functioning including selective attention, memory, executive function, and global clinical rating

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Director — Novartis Pharmaceuticals